CLINICAL TRIAL: NCT03655392
Title: Clinical, Functional and Inflammatory Evaluation in Asthmatic Patients After a Simple Short-Term Educational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other); Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Beatriz Mangueira Saraiva Romanholo, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IAMSPE
Record Dates: First submitted 2018-03-28; First posted 2018-08-31 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Asthma; Inflammation; Patient Relations, Nurse; Spirometry
Keywords: asthma; inflammation; patients education; spirometry
MeSH Terms: conditions — Asthma; Inflammation | interventions — Spirometry; Respiratory Function Tests; Peak Expiratory Flow Rate

STUDY DESIGN:
Intervention Model Description: 64 adult asthmatic patients (18-70 years old) were randomized into two groups: intervention group (IG) (n=38) or control group (CG) (n=26). IG patients were submitted to three 30-minutes intervention of a shortterm educational program delivered by a nurse at 3 mensal intervals. CG group did not receive educational intervention. All patients were submitted to a spirometry, induced sputum collection, nitric oxide measure, collecting exhaled condensed (cytokine analysis) air and it's ph measure, Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality Life Questionnaire (AQLQ), Beck Depression Inventory (BDI), and answered a symptoms diary, Statistical analysis: repeated measures (Sigma Plot Software 3.0).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 64 adult asthmatic patients (18-70 years old) were randomized into two groups: intervention group (IG) (n=38) or control group (CG) (n=26). IG patients were submitted to a individualized educational program: three 30-minutes intervention of a shortterm educational program delivered by a nurse at 3 monthly visits. CG group did not receive educational intervention. All patients were submitted to a spirometry, induced sputum collection, nitric oxide measure, exhaled breath condensate air measurement, and answered the questionnaires ACT, ACQ, AQLQ, BDI: Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality Life Questionnaire (AQLQ), Beck Depression Inventory (BDI). All participants also answered a symptoms diary about asthma symptoms and peak flow measure.
  Interventions: Behavioral: Individualized educational program; Diagnostic Test: Induced sputum collection; Diagnostic Test: Spirometry; Diagnostic Test: Nitric oxide measure; Other: Questionnaires ACT, ACQ, AQLQ, BDI; Other: Symptoms Diary; Diagnostic Test: Peak flow measure; Diagnostic Test: Exhaled breath condensate air measurement
- Control Group (Experimental): 64 adult asthmatic patients (18-70 years old) were randomized into two groups: intervention group (IG) (n=38) or control group (CG) (n=26). IG patients were submitted to three 30-minutes intervention of a shortterm educational program delivered by a nurse at 3 montly visits. CG group did not receive educational intervention. All patients were submitted to a spirometry, induced sputum collection, nitric oxide measure, exhaled breath condensate air measurement, and answered the questionnaires: Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality Life Questionnaire (AQLQ), Beck Depression Inventory (BDI). All participants also answered a symptoms diary about asthma symptoms and peak flow measure.
  Interventions: Diagnostic Test: Induced sputum collection; Diagnostic Test: Spirometry; Diagnostic Test: Nitric oxide measure; Other: Questionnaires ACT, ACQ, AQLQ, BDI; Other: Symptoms Diary; Diagnostic Test: Peak flow measure; Diagnostic Test: Exhaled breath condensate air measurement

INTERVENTIONS:
Behavioral: Individualized educational program — IG patients were submitted to three 30-minutes intervention of a individualized shortterm educational program delivered by a nurse, were given explanations about general aspects of the disease, prevention methods and about the importance and correct use of inhaled corticosteroids, with an educational video showing the use of the device
  Other Names: Short term educational program
  Arms: Intervention Group
Diagnostic Test: Induced sputum collection — All participants performed induced sputum collection
  Other Names: Induced sputum
Diagnostic Test: Spirometry — All participants performed spirometry test using a Koko spirometer. Pulmonary function was assessed by spirometry prebronchodilator, after withholding short-acting beta-agonists for ≥ 6 hours and long-acting beta-agonist for ≥ 24hours. Forced expiratory volume in one second (FEV1) % predicted was used as a proxy variable for overall lung function.
  Other Names: Lung function test
Diagnostic Test: Nitric oxide measure — All participants performed nitric oxide measure in three Mylar bags and measure was performed in a NOA280 Sievers equipment. For collection the patients blew in the balloons through a sterile nozzle in the equipment collector without prejudice or damage to the patient.
  Other Names: NO measure
Other: Questionnaires ACT, ACQ, AQLQ, BDI — All participants answered standardized questionnaires about asthma symptoms and depression: Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality Life Questionnaire (AQLQ), Beck Depression Inventory (BDI)
Other: Symptoms Diary — All participants were instructed to note in the morning and evening before the use of routine inhaled corticosteroids, asthma symptoms (coughing, wheezing, shortness of breath, use of emergency inhaled corticosteroids) and three measures of peak expiratory flow (individual, provided to patients) and to return this completed diary at each study visit
Diagnostic Test: Peak flow measure — All participants registered three peak flow measures in the symptoms diary by morning and night before the use of routine inhaled corticosteroids. Peak flow was measured by the electronic peak flow meter (Mini-Wright).
  Other Names: Peak flow
Diagnostic Test: Exhaled breath condensate air measurement — Exhaled breath condensate was collect during 15 to 20 minutes in a Turbo DECCS equipment (Medivac SRL, Italy) in a sterile buccal of the own apparatus with the aid of a nasal clip with the participant breathing normally without any effort or damage.
  Other Names: EBC collection

SUMMARY:
Background: Patient education is one of the pillars of asthma treatment according to GINA guidelines. It has considered essential for adherence to treatment and for correct technique of inhaled devices.

DETAILED DESCRIPTION:
Objective: analyze clinical, functional and inflammatory features of adult patients with partly controlled and uncontrolled asthma, before and after an educational intervention. Methods: 58 adult asthmatic patients (18-70 years old) were randomized into two groups: intervention group (IG) (n=38) or control group (CG) (n=26). IG patients were submitted to three 30-minutes intervention of a shortterm educational program delivered by a nurse in 3 visits with a one-month interval. CG group did not receive educational intervention. All patients were submitted to a spirometry, induced sputum collection, nitric oxide measure, collecting exhaled condensed (cytokine analysis) air and it's ph measure, Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality Life Questionnaire (AQLQ), Beck Depression Inventory (BDI), and answered a symptoms diary, Statistical analysis: repeated measures (Sigma Plot Software 3.0).

ELIGIBILITY:
Inclusion criteria:

* Non-smokers or those who stopped smoking more than five years ago
* Age between 18-69 years
* Be legally capable
* Response to the short-acting bronchodilator FEV1> 12% and> 200 mL
* Absence of upper airway infection during 30 days and associated systemic diseases

Exclusion criteria:

* Smokers
* Over 70 years old
* Airway infection
* Legally incapable persons
* Diseases that may affect respiratory function

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Induced sputum samples to assess airway inflammation | One day
  Induced sputum samples were collected in 3 visits with a one-month interval to assess the degree of airway inflammation. Markers of inflammation included eosinophils, neutrophils, macrophages, lymphocytes and total cell counts, as well as cytokines in the sputum supernatant. In the processing performed the subjects received up to three nebulizations with 3% hypertonic saline, the aerosol was generated by an ultrasonic nebulizer (Ultraneb 99; DeVilbiss, Somerset, PA) each challenge was monitored with peak flow before, after and between nebulizations.
Pulmonary function by spirometry | One day
  Pulmonary function was assessed by spirometry pre and after bronchodilator (Salbutamol, short action beta-agonist), according to ATS guidelines, in 3 visits with a one-month interval after withholding short-acting beta-agonists for ≥ 6 hours and long-acting betaagonist for ≥ 24hours. Forced expiratory volume in one second (FEV1) % predicted was used as a proxy variable for overall lung function
Asthma control by Asthma Control Test (ACT) | One day
  Asthma Control Test (ACT) was used to assess clinical control of asthma in the last month; is a questionnaire composed of five questions (score varying from 5 to 25 points) assessing asthma in relation to physical activity limitation, nocturnal and diurnal symptoms, shortness of breath and use of rescue medication. The higher the overall score, the greater the asthma control, and a 3-point difference in the mean ACT score is considered a clinically relevant change.
Depression symptoms by Beck Depression Inventory II (BDI II) | One day
  To evaluate the symptoms of depression reported in the last 30 days, BDI II was used, a questionnaire composed of 21 items with scores ranging from 0 to 63 points, the higher the score the worse the severity of the symptoms
Asthma quality of life by Asthma Quality of Life Questionnaire (AQLQ) | One day
  Asthma quality of life was assessed using the AQLQ, which has four domains: activity limitations, symptoms, emotional function and environmental stimuli. A higher AQLQ score indicates a better quality of life.
Fractional exhaled nitric oxide (FeNO) | One day
  FeNO was collected also to assess airway inflammation in acoordance with the ATS recommendations; all measurements were determinad by chemiluminscence (Sievers 280). This analysis procedure was performed by a blinded investigator. The patients were advised to blow into a Mylar bag, with a breath pressure of 12 cmH20, monitored by the pressure gauge, reaching a flow rate of 200 mL/s.
Exhaled breath condensate (EBC) | One day
  A Turbo DECCS® condenser (Medivac SRL, Italy) (29) was used which was cooled to -20øC for at least thirty minutes prior to use. The subjects were instructed to perform oral breathing using the mouthpiece of the equipment and with the aid of a nasal clip. The EBC (exhaled breath condensate) was collected for 15 to 20 minutes in tidal volume for pH analysis and cytokine dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Soraia N Felix, Master, Principal Investigator — IAMPSE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felix SN, Agondi RC, Aun MV, Olivo CR, de Almeida FM, Amorim TS, Cezario JC, Giavina-Bianchi P, Tiberio IFLC, de Martins MA, Romanholo BMS. Clinical, functional and inflammatory evaluation in asthmatic patients after a simple short-term educational program: a randomized trial. Sci Rep. 2021 Sep 14;11(1):18267. doi: 10.1038/s41598-021-97846-8. PMID 34521963